CLINICAL TRIAL: NCT04898205
Title: Cardiopulmonary Rehabilitation in COVID-19 Longhaulers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Noah Greenspan (Other)
Collaborators: University of Dayton (Other)
Responsible Party: Sponsor-Investigator, Noah Greenspan, Founder, Pulmonary Wellness Foundation
Organization: Pulmonary Wellness Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PLM UD 2021
Record Dates: First submitted 2021-05-17; First posted 2021-05-24 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Viral Syndrome
Keywords: Post-COVID Syndrome; Post-acute COVID; Long COVID
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: This study entails 24 treatment sessions. The first 8 sessions involve four experimental conditions: 1) exercise + oxygen (treatment), exercise + air (active control), oxygen only (active control), air only (placebo). Pre-treatment testing will then be repeated, after which all participants will crossover to 16 sessions of exercise + oxygen.
Who Masked: Participant
Masking Description: All participants will be blind to whether they receive supplemental oxygen or air during the first 8 sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treadmill Exercise with Supplemental Oxygen (Experimental): Participants will receive 24 sessions (2 x week for 12 weeks) of treadmill exercise combined with 6 liters per minute of supplemental oxygen via nasal cannula during exercise and 5-minutes of recovery. The first treadmill session will last 25% longer than the exercise tolerance test, but at a lower intensity, such that 80-100% of peak exercise intensity calculated from the exercise tolerance test MET is achieved within three sessions, after which time and intensity will be increased by no more than 0.5 METS, as tolerated based on symptoms and vitals. Heart rate, rhythm, and oxygen saturation will be continuously monitored, and blood pressure readings will be obtained every three to five minutes.
  Interventions: Other: Treadmill Exercise; Other: Concentrated Oxygen
- Treadmill Exercise with Air (Sham Comparator): Participants will receive 8 sessions (2 x week for 4 weeks) of treadmill exercise combined with air delivered via nasal cannula during exercise and 5-minutes of recovery. They will then cross-over to 16 sessions of treadmill exercise combined with 6 liters per minute of supplemental oxygen via nasal cannula during exercise and 5-minutes of recovery. The first treadmill session will last 25% longer than the exercise tolerance test, but at a lower intensity, such that 80-100% of peak exercise intensity calculated from the exercise tolerance test MET is achieved within three sessions, after which time and intensity will be increased by no more than 0.5 METS, as tolerated based on symptoms and vitals. Heart rate, rhythm, and oxygen saturation will be continuously monitored, and blood pressure readings will be obtained every three to five minutes.
  Interventions: Other: Treadmill Exercise; Other: Concentrated Oxygen; Other: Concentrated Air
- Supplemental Oxygen Only (Sham Comparator): Participants will receive 8 treatment sessions (2 x week for 4 weeks) of 6 liters per minute of continuous oxygen via nasal cannula for 30 minutes at rest. Heart rate, rhythm, and oxygen saturation will be continuously monitored, and blood pressure readings will be obtained every three minutes. They will then cross-over to 16 sessions of treadmill exercise combined with 6 liters per minute of supplemental oxygen via nasal cannula during exercise and 5-minutes of recovery. The first treadmill session will last 25% longer than the exercise tolerance test, but at a lower intensity, such that 80-100% of peak exercise intensity calculated from the exercise tolerance test MET is achieved within three sessions, after which time and intensity will be increased by no more than 0.5 METS, as tolerated based on symptoms and vitals. Heart rate, rhythm, and oxygen saturation will be continuously monitored, and blood pressure readings will be obtained every three to five minutes.
  Interventions: Other: Treadmill Exercise; Other: Concentrated Oxygen
- No Intervention (Placebo Comparator): Participants will receive 8 treatment sessions (2 x week for 4 weeks) of air via nasal cannula for 30 minutes at rest. Heart rate, rhythm, and oxygen saturation will be continuously monitored, and blood pressure readings will be obtained every three minutes. They will then cross-over to 16 sessions of treadmill exercise combined with 6 liters per minute of supplemental oxygen via nasal cannula during exercise and 5-minutes of recovery. The first treadmill session will last 25% longer than the exercise tolerance test, but at a lower intensity, such that 80-100% of peak exercise intensity calculated from the exercise tolerance test MET is achieved within three sessions, after which time and intensity will be increased by no more than 0.5 METS, as tolerated based on symptoms and vitals. Heart rate, rhythm, and oxygen saturation will be continuously monitored, and blood pressure readings will be obtained every three to five minutes.
  Interventions: Other: Treadmill Exercise; Other: Concentrated Oxygen; Other: Concentrated Air

INTERVENTIONS:
Other: Treadmill Exercise — The cardiopulmonary rehabilitation protocol utilizes progressive treadmill exercise with alternating increases in intensity and incline with no more than 0.5 Met increase per session.
  Other Names: Supplemental oxygen (6 liters per minute)
Other: Concentrated Oxygen — Supplemental oxygen from a concentrator (6 liters per minute) will be provided via nasal cannula regardless of oxygen saturation.
Other: Concentrated Air — Room air will be delivered through an concentrator provided via nasal cannula.
  Arms: No Intervention; Treadmill Exercise with Air

SUMMARY:
This study will test the efficacy of treadmill exercise combined with supplemental oxygen during exercise and recovery for the treatment of persistent post-acute COVID-19 symptoms. Participants will be pseudo-randomized (stratified by age) to one of four conditions for 8 treatment sessions: 1) treadmill exercise plus supplemental oxygen, 2) treadmill exercise plus air, 3) supplemental oxygen only, 4) air only. All participants will then cross-over and receive 16 additional sessions of treadmill exercise plus supplemental oxygen.

DETAILED DESCRIPTION:
This study will test the efficacy of a COVID-19 specific cardiopulmonary rehabilitation protocol for treatment of persistent post-acute COVID symptoms and to study the impact of cardiopulmonary improvement on cognition, mental health, and function. Participants (N=36) with persistent post-acute COVID symptoms will undergo pre-treatment neurocognitive, orthostatic tolerance, and exercise tolerance tests before being pseudo-randomized (stratified by age and sex) to one of four conditions (all of which occur twice a week): 1) 8 sessions of treadmill exercise plus supplemental oxygen, 2) 8 sessions of treadmill exercise plus air, 3) 8 sessions of supplemental oxygen only, and 4) 8 sessions of air only. The pre-treatment testing will be repeated, after which all participants will receive 16 additional sessions of treadmill exercise plus supplemental oxygen, followed by post-treatment testing. All participants will complete baseline measures of physical and mental health, physical function, emotional wellbeing, and coping. A brief symptom measure will be collected daily and physical function, mental health, and emotional wellbeing will be assessed weekly.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-60
* Contracted COVID-19 between February - July 2020
* Has been clinician-diagnosed with COVID-19 based on PCR/antigen testing, antibody testing, or clinical symptoms
* Is currently experiencing one or more of the following symptoms, which began only after contracting COVID-19 : dyspnea, cough, chest pain, tachycardia or other arrhythmias, hypertension, hypotension, blood pressure lability, oxygen desaturation, exercise/activity intolerance, fatigue, or dizziness.
* Has been cleared by a physician for exercise and supplemental oxygen.
* Has the capacity to provide written, informed consent
* Able to complete questionnaires in English

Exclusion Criteria:

* History of any of the following per the American College of Sports Medicine exercise testing guidelines (American College of Sports Medicine et al., 2018) to be determined during a screening consultation:

  1. Acute myocardial infarction within the past two days
  2. Ongoing unstable angina
  3. Uncontrolled cardiac arrhythmias
  4. Active endocarditis
  5. Symptomatic severe aortic stenosis
  6. Decompensated heart failure
  7. Active pulmonary embolism, pulmonary infarction, or deep venous thrombosis
  8. Active myocarditis or pericarditis
  9. Acute aortic dissection
  10. Physical disability that precludes safe and adequate testing
* Participants who demonstrate orthostatic intolerance or oxygen desaturation (<90%) during the exercise tolerance test will no longer be eligible for the study because it is not safe for them to exercise on a treadmill.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-01-20 (Estimated); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
Heart rate and rhythm response to exercise and positional changes | Up to 24-weeks
  Heart rate and rhythm will be measured using 3-lead ECG telemetry
Blood pressure response to exercise and positional changes | Up to 24-weeks
  Blood pressure will be measured via manual cuff
Activity metabolic equivalent of task (MET) tolerated | Up to 24-weeks
  MET will be computed based upon peak exercise speed (MPH) and incline % gradation). Scores are expected to range from 1.8 to 12.1 (but can be higher is speed exceeds 3.9 MPH). Higher METs indicate more energy output.
Breathlessness | Up to 24-weeks
  Breathlessness will be assessed during peak exercise via self-report using the Borg Dyspnea scale. Scores can range from 0 to 20 and higher scores indicate more breathlessness
Rate of perceived exertion (RPE) | Up to 24-weeks
  RPE will be assessed during peak exercise via self-report using the Borg RPE scale. Scores can range from 0 to 20 and higher scores indicate more RPE.
Cognition (attention, short, delayed, and working memory, verbal fluency, and abstraction). | Up to 24-weeks
  Cognition will be assessed with the Repeatable Battery for the Assessment of Neuropsychological Status Update (RBANS-U) List Learning, List Recall, List Recognition, Story Memory, Story Recall, Semantic Fluency and Picture Naming subtests and the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) Similarities and Digit Span subtests. All scores will be standard scores based on age norms.
Post-acute COVID symptoms (PACS) | Up to 24-weeks
  Frequency and severity of 38 PACS symptoms will be assessed daily via an online survey. Each symptom will be rated on a scale of 0 (not present) to 5 (severe).
Physical Function | Up to 24-weeks
  Physical function will be measured weekly via self-report with the Physical Function Short Form-36. Scores can range from 0 to 100 and higher scores indicate better function.

SECONDARY OUTCOMES:
Depression | Up to 24-weeks
  Depression will be measured weekly with the Center for Epidemiological Studies Depression Scale - Revised (CESD-R). Scores range from 0 to 60 and higher scores indicate greater depression severity.
Generalized anxiety | Up to 24-weeks
  Generalized anxiety will be measured weekly using the Generalized Anxiety Disorder - 2 (GAD-2). Scores range from 0 to 6 and higher scores indicate greater anxiety severity.
State anxiety | Up to 24-weeks
  Anxiety will be measured weekly using the State Trait Anxiety Inventory (STAI) - State scale. Scale scores range from 20 to 80, with higher scores indicating greater state anxiety.
Trait anxiety | Up to 24-weeks
  Trait anxiety will be measured weekly using the State Trait Anxiety Inventory (STAI) - Trait scale. Scores can range from 20 to 80, with higher scores indicating greater trait anxiety.
Improvement in quality of life | Up to 24-weeks
  Quality of life will be measured weekly with the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF). Raw scores range from 14 to 70 and will be converted to a percentage score based on the following formula:
  (raw total score -minimum score)/(maximum possible raw score -minimum score). Higher scores indicate greater life satisfaction.
Perception of cognitive function | Up to 24-weeks
  Perception of cognitive function will be assessed with the Neuro-QOL Cognitive function subscale which measures self-reported cognitive functioning over the past week, including perceptions of memory, executive functions, processing speed, and learning. Raw scores can range from 8 to 40, and will be converted to T-scores based on the administration manual norms. Higher scores indicated better perceived cognitive function.
  We have modified the baseline administration to also assess whether perceived cognitive function has changed since onset of acute COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Greenspan, DPT, Principal Investigator — Pulmonary Wellness Foundation; Julie Walsh-Messinger, Ph.D., Principal Investigator — University of Dayton
Locations (1):
- Post-COVID Rehabilitation and Recovery Clinic at H&D Physical Therapy, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Upon conclusion of the study, we will share de-identified data upon request.

REFERENCES:
- See also: Pulmonary Wellness Foundation — https://pulmonarywellness.org/research/
- See also: Pulmonary Wellness Post-COVID Rehabilitation and Recovery Clinic at H&D Physical Therapy — https://www.hdphysicaltherapy.com/post-covid/
- See also: Psychopathology, Personality, and Affective Science (PPAS) Laboratory at the University of Dayton — https://juliewalshmessinger.weebly.com/research-studies.html